CLINICAL TRIAL: NCT06127316
Title: The Effects of Heel Distraction Height on Foot Loading With Carbon Fiber Custom Dynamic Orthoses
Acronym: CDODistract
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Fabtech Systems (Unknown)
Responsible Party: Principal Investigator, Jason Wilken, Associate Professor, University of Iowa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 202302397; CDMRP-OP230037 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Traumatic Lower Limb Injury
Keywords: Plantar Force; Ankle Foot Orthosis; Carbon Fiber Orthosis; Biomechanics

STUDY DESIGN:
Intervention Model Description: In this study, forces acting under the foot (hindfoot, midfoot, forefoot, and total foot) will be measured using wireless Loadsol insoles (Novel GMBH, St. Paul, MN) as participants walk without an orthosis (NoCDO) and with a CDO with three different posterior strut lengths resulting in three different levels of heel distraction (0cm, 1cm, 2cm) at self-selected and controlled speeds. Gait kinematics and kinetics will be measured using infra-red motion capture cameras (Vicon Motion Systems Ltd., Denver, CO) and force plates (AMTI, Watertown, MA). Testing order of the CDO conditions will be randomized to prevent influence of testing order.
Who Masked: Participant
Masking Description: Participants will be blinded, to the greatest extent possible, to the different CDO heel distraction heights.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- NoCDO (No Intervention): Participants will complete study activities without a CDO
- 0cm Distraction (Experimental): Participants will complete study activities while wearing a CDO with 0cm of heel distraction height
  Interventions: Device: Carbon Fiber Custom Dynamic Orthosis (CDO)
- 1cm Distraction (Experimental): Participants will complete study activities while wearing a CDO with 1cm of heel distraction height
  Interventions: Device: Carbon Fiber Custom Dynamic Orthosis (CDO)
- 2cm Distraction (Experimental): Participants will complete study activities while wearing a CDO with 2cm of heel distraction height
  Interventions: Device: Carbon Fiber Custom Dynamic Orthosis (CDO)

INTERVENTIONS:
Device: Carbon Fiber Custom Dynamic Orthosis (CDO) — The carbon fiber custom dynamic orthoses (CDOs) used in this study will consist of a semi-rigid carbon fiber footplate, a carbon fiber posterior strut, and a proximal cuff that wraps around the leg below the knee. The CDO will be modular in design which will allow three carbon fiber struts of the same stiffness and differing lengths to be used to implement 0cm, 1cm, and 2cm levels of heel distraction height. A longer posterior strut will move the carbon fiber footplate away from the participants foot to create the heel distraction height.
  Other Names: Ankle Foot Orthosis (AFO)
  Arms: 0cm Distraction; 1cm Distraction; 2cm Distraction

SUMMARY:
Carbon fiber custom dynamic orthoses (CDOs) and unloading ankle foot orthoses (AFOs) have shown varying levels of success in reducing forces acting on different regions of the bottom of the foot during gait. CDOs and unloading AFOs have shown differing offloading capabilities across different regions of the foots (hindfoot, midfoot, forefoot) which may be related to a distinct difference between CDOs and unloading AFOs: CDOs do not suspend, or distract, the foot away from the footplate. The purpose of this study is to determine the effects of CDOs and heel distraction height (the distance between the heel and the footplate) on limb loading and motion during gait as well as patient reported pain, and comfort.

DETAILED DESCRIPTION:
Carbon fiber custom dynamic orthoses (CDOs) have been used to improve function, reduce pain, and offload the foot and ankle for individuals with a number of conditions affecting the lower extremity. CDOs consist of a proximal cuff that wraps around the leg just below the knee, a posterior carbon fiber strut that bends to store and return energy during mid to late stance, a semi-rigid carbon fiber footplate, and, in some cases, a foam heel wedge placed in the shoe. Unloading ankle foot orthoses (AFOs) have also been used for a number of lower extremity conditions, including traumatic injuries, in effort to reduce forces and pressure acting under the foot. Unloading AFOs have been created using many different designs, which include a proximal cuff just below the knee, a rigid strut (made of metal, plastic, etc.), and some sort of foot component (footplate, shoe, etc.).

Both CDOs and unloading AFOs have shown varying levels of success in reducing forces acting on different regions of the bottom of the foot during gait. The differences in loading may be related to a distinct difference between CDOs and unloading AFOs: CDOs do not suspend, or distract, the foot away from the footplate.

The purpose of this study is to determine the effects of CDOs and heel distraction height (the distance between the heel and the footplate) on limb loading and motion as well as patient reported pain and comfort. In this study, forces acting under the foot will be measured using wireless Loadsol insoles (Novel GMBH, St. Paul, MN) as participants walk without an orthosis (NoCDO) and with a CDO with three different posterior strut lengths resulting in three different levels of heel distraction (0cm, 1cm, 2cm) at self-selected and controlled speeds. Additionally, gait kinematic and kinetics will be measured using infrared motion capture cameras (Vicon Motion Systems Ltd., Denver, CO) and force plates (AMTI, Watertown, MA). Participants will be provided a lift for the contralateral limb to reduce the effects of leg length discrepancies during walking. Loadpad force measuring sensors (Novel GMBH, St. Paul, MN) will be used to measure forces within the CDO proximal cuff. After walking in each condition, participants will complete questionnaires concerning pain and orthosis comfort.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-65 years
2. Traumatic hindfoot injury (soft tissue injury or fracture affecting the hindfoot or ankle)
3. Mechanical pain with limb loading (>=4/10 on Numerical Pain Rating Scale)
4. Ability to walk 50 feet at a slow to moderate pace
5. Ability to walk without a cane or crutch
6. Ability to read and write in English and provide written informed consent

Exclusion Criteria:

1. Diagnosis with a moderate or severe brain injury
2. Diagnosis with a physical or psychological condition that would preclude functional testing (e.g., cardiac condition, clotting disorder, pulmonary condition, etc.
3. Ankle weakness resulting from spinal cord injury or central nervous system pathology
4. Nerve, muscle, bone, or other condition limiting function in the contralateral extremity
5. Rheumatoid or inflammatory arthritis
6. Necrosis of any bones in the foot or ankle
7. Pain of 8/10 or greater during walking
8. Uncorrected visual or hearing impairments
9. Require use of a knee stabilizing device to perform daily activities (i.e., Knee ankle foot orthosis, knee orthosis, etc.)
10. Pregnancy
11. Body mass index greater than 40 kg/m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Peak Force (forefoot) | Baseline
  Plantar forces (N) will be measured across the forefoot (distal 40% of sensor) as participants walk without a CDO and with each CDO.
Force Impulse (forefoot) | Baseline
  Plantar force impulse (Ns) across the forefoot (distal 40% of sensor) will be calculated using the integral of the force over the stance phase as participants walk without a CDO and with each CDO.
Peak Force (hindfoot) | Baseline
  Plantar forces (N) will be measured across the hindfoot (proximal 30% sensor) as participants walk without a CDO and with each CDO.
Force Impulse (hindfoot) | Baseline
  Plantar force impulse (Ns) across the hindfoot (proximal 30% sensor) will be calculated using the integral of the force over the stance phase as participants walk without a CDO and with each CDO.
Numerical Pain Rating Scale | Baseline
  Pain will be assessed using a standard 11-point numerical pain rating scale, in which 0 = no pain and 10 = worst pain imaginable
Modified Socket Comfort Score | Baseline
  Comfort scores range from 0 = most uncomfortable to 10 = most comfortable, and from 0 = least smooth to 10 = most smooth

SECONDARY OUTCOMES:
Peak Force (total foot) | Baseline
  Plantar forces (N) will be measured across the total foot (100% of sensors) as participants walk without a CDO and with each CDO.
Force Impulse (total foot) | Baseline
  Plantar force impulse (Ns) across the total foot (100% of sensors) will be calculated using the integral of the force over the stance phase as participants walk without a CDO and with each CDO.
Peak Force (midfoot) | Baseline
  Plantar forces (N) will be measured across the midfoot (middle 30% of sensor) as participants walk without a CDO and with each CDO.
Force Impulse (midfoot) | Baseline
  Plantar force impulse (Ns) across the midfoot (middle 30% of sensor) will be calculated using the integral of the force over the stance phase as participants walk without a CDO and with each CDO.
Ankle Range of Motion | Baseline
  Peak ankle dorsiflexion (degrees) during gait.
Peak Ankle Moment | Baseline
  Peak ankle plantarflexion moment (Nm/kg) during gait.
Peak Ankle Power | Baseline
  Peak ankle push-off power (W/kg) during gait.

OTHER OUTCOMES:
Semi-Structured Interview | Baseline
  Participants will be asked a number of open ended questions to help determine what factors influenced their perception of each study condition.

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Wilken, PT,PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT06127316/Prot_SAP_000.pdf